CLINICAL TRIAL: NCT00167271
Title: Efficacy of Computer and SenseWear Technologies for Promoting Health in People With Fibromyalgia: A Randomized Clinical Trial
Brief Title: Promoting Health in People With Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: U.S. Department of Education (U.S. Federal Agency)
Responsible Party: Joan C. Rogers, PhD, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 020771
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2011-02-21 (Estimated); Status verified 2011-02

CONDITIONS: Fibromyalgia
Keywords: Cognitive therapy
MeSH Terms: conditions — Fibromyalgia | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental (Experimental): Computerized cognitive, behavioral therapy with Body Media armband to collect data about activity, which subjects could review each evening.
  Interventions: Behavioral: Cognitive Behavior Therapy
- Control (Active Comparator): Subjects given pamphlets from the Arthritis Foundation
  Interventions: Behavioral: Cognitive Behavior Therapy

INTERVENTIONS:
Behavioral: Cognitive Behavior Therapy — Experimental: Computerized cognitive, behavioral therapy with Body Media armband to collect data about activity, which subjects could review each evening.
  Other Names: Control

SUMMARY:
Body worn sensors and the Internet can be used to self-monitor daily behavior and promote a healthier lifestyle in women with fibromyalgia.

DETAILED DESCRIPTION:
Fibromyalgia is among the most common diffuse pain syndromes, affecting about 1 of every 10 rheumatology patients. People with fibromyalgia experience widespread chronic pain and fatigue that negatively influences their activity participation (causes disability) and overall quality of life.

The purpose of this 3-year study is to use a cognitive-behavioral intervention to facilitate adoption of a wellness lifestyle in people with fibromyalgia. Specifically, we will test the efficacy of a health promotion computer program (Balance Center) used in conjunction with a wearable sensor (SenseWearTM) for developing a wellness lifestyle and improving the quality of life of adults with fibromyalgia. Balance Center software is a health promotion computer program that helps consumers to: (1) establish goals in the areas of physical activity, nutrition, participation in meaningful, productive activities, sleep, stress-reducing activities, and emotional state; (2) monitor progress toward established goals; and, (3) assess the relationship between these areas in one's daily life. In addition, based on consumer input, it offers suggestions for developing a wellness lifestyle. SenseWearTM, provides objective data about activity level and stress level for consumers to use in combination with the self-assessment data provided by the Balance Center.

In this randomized controlled clinical trial, the Experimental (Balance Center + SenseWearTM) Intervention is compared to a Usual Care, control group. Seventy-two adults (36 = Experimental; 36 = Control) with fibromyalgia will be randomized and followed for 6 weeks, exclusive of Baseline and Posttesting. The hypotheses to be tested are: Participants randomized to the Experimental Condition will demonstrate significantly (a) more physical activity, (b) a healthier, wellness lifestyle, and (c) fewer symptoms of fibromyalgia. In addition, the relationship between the decrease in fibromyalgia-related impairment on daily life and physical activity and a wellness lifestyle will be stronger at Posttesting than at Baseline in the Experimental Group, compared to the Control Group. The anticipated outcome of the intervention is more effective self-management of lifestyle and symptoms so that one can "live well with fibromyalgia."

ELIGIBILITY:
Inclusion Criteria:

* be at least 18 years of age
* meet the American College of Rheumatology criteria for fibromyalgia
* diagnosed with fibromyalgia at least 1 year prior to admission to the study
* have sufficient vision to operate a computer
* be English speaking
* have a private telephone line

Exclusion Criteria:

* live beyond a 40 mile radius of Pittsburgh

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2002-10; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Fibromyalgia Impact Questionnaire, symptom reduction | 6 weeks
  Queries about symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Joan C. Rogers, Ph.D., Principal Investigator — University of Pittsburgh
Locations (1):
- Subjects' homes, Pittsburgh, Pennsylvania, United States